CLINICAL TRIAL: NCT03555630
Title: Effect of Age on Reference Values for Thromboelastography in Pregnant Women With Pre-eclampsia
Brief Title: Thromboelastogram in Postdelivery Preeclamptic Patients
Status: Completed | Type: Observational
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Efrain Riveros Perez, MD, Assistant Professor Department of Anesthesiology and Perioperative Medicine, Augusta University
Other Study IDs: [1167446
Record Dates: First submitted 2018-06-01; First posted 2018-06-13 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Preeclampsia; Coagulation Disorder; Pregnancy Complications
MeSH Terms: conditions — Pre-Eclampsia; Hemostatic Disorders; Pregnancy Complications | interventions — Thrombelastography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Post-cesarean preeclampsia
  Interventions: Diagnostic Test: Thromboelastogram
- Post spontaneous vaginal delivery preeclampsia
  Interventions: Diagnostic Test: Thromboelastogram

INTERVENTIONS:
Diagnostic Test: Thromboelastogram — Blood sample processing for thromboelastogram

SUMMARY:
There are no studies evaluating the effect of aging on hemostasis of preeclamptic patients. Additionally, although there are some studies that establish normal reference values for TEG profiles in healthy term pregnant patients, conflicting results have been found in preeclampsia. Reference values are important to establish baseline parameters in cases of pre-eclampsia complicated by postpartum hemorrhage. The investigators will evaluate reference values for TEG in postdelivery preeclamptic patients and the difference between vaginal delivery and cesarean section.

DETAILED DESCRIPTION:
After approval by the Institutional Review Board and informed consent from participants, the investigators are obtaining blood samples for TEG processing, from pregnant patients admitted to the maternity unit of Augusta University Medical Center. Patients are being classified in 2 groups: term pregnant patients with diagnosis of pre-eclampsia who undergo cesarean section and those having spontaneous vaginal delivery. Each group will be divided into subgroups according to maternal age: 18-25 years, 26-35 years, >36 years. Pre-eclampsia is defined and classified according to the definitions of the American College of Obstetricians and Gynecologists published in 2013.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years Mental competence Gestational age > 37-week Informed consent Diagnosis of preeclampsia (with or without features of severity)

Exclusion Criteria:

Gestational age < 37-week Known bleeding or thrombotic diathesis Use of aspirin or unfractionated or low-molecular weight heparin within the last 48 hours BMI > 35 Maternal comorbid conditions other than preeclampsia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant patients
Study Population: Term pregnant patients with preeclampsia
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
R time | 10 minutes
  Reaction time of whole blood

SECONDARY OUTCOMES:
K time | 10 minutes
  Activation time
Maximum amplitude | 10 minutes
  Amplitude in relation to platelet count and function
LY-30 | 30 minutes
  Lysis at 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No